CLINICAL TRIAL: NCT04562558
Title: A Prospective，Multicenter，Randomized Trial of Biweekly Single-dose Actinomycin-D Versus Multi-day Methotrexate Protocol for the Treatment of Low-risk Gestational Trophoblastic Neoplasia
Brief Title: Biweekly Actinomycin-D Treatment or Multi-day Methotrexate Protocol in Low-risk Gestational Trophoblastic Neoplasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: xiang yang (Other)
Responsible Party: Sponsor-Investigator, xiang yang, the Director of Gynecological Oncology Center at Peking Union Medical College Hospital, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-LRGTN-SINGLE DRUG-0222
Record Dates: First submitted 2020-09-13; First posted 2020-09-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gestational Trophoblastic Tumor; Gestational Trophoblastic Neoplasia; Stage I Gestational Trophoblastic Tumor; Stage II Gestational Trophoblastic Tumor; Stage III Gestational Trophoblastic Tumor; Invasive Mole; Choriocarcinoma
Keywords: gestational trophoblastic neoplasia; actinomycin-D; methotrexate; low-risk
MeSH Terms: conditions — Gestational Trophoblastic Disease; Hydatidiform Mole, Invasive; Choriocarcinoma | interventions — Methotrexate; Leucovorin; Dactinomycin

STUDY DESIGN:
Intervention Model Description: A prospective，multicenter，randomized trial with two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1-Methotrexate (Experimental): Patients receive methotrexate intramuscularly（50mg） on Days 1, 3, 5, 7 (4 doses per cycle) with Leucovorin (15mg) on Days 2, 4, 6, 8. Repeat every 14 days. Patients continue on treatment until beta HCG titer is below the institutional normal. Patients then receive 2-3 additional consolidation treatment. If the level of hCG become stationary for at least 2 course of single-agent chemotherapy or rise again, the patient will be referred to multi-course chemotherapy. FAV regimen is preferred, or EMA-CO regimen can also be selected if FAV is unavailable.
  Interventions: Drug: Methotrexate; Drug: Leucovorin
- Arm 2-Dactinomycin (Experimental): Patients will receive IV pulse actinomycin-D (1.25mg/m2，2mg max dos) every 14 days. Patients continue on treatment until beta HCG titer is below the institutional normal. Patients then receive 2-3 additional consolidation treatment.If the level of hCG become stationary for at least 2 course of single-agent chemotherapy or rise again, the patient will be referred to multi-course chemotherapy. FAV regimen is preferred, or EMA-CO regimen can also be selected if FAV is unavailable.
  Interventions: Drug: Dactinomycin

INTERVENTIONS:
Drug: Methotrexate — 50mg intramuscularly on Days 1, 3, 5, 7 . Repeat every 14 days
  Other Names: MTX
  Arms: Arm1-Methotrexate
Drug: Leucovorin — 15mg intramuscularly on Days 2, 4, 6, 8. Repeat every 14 days
  Other Names: Calcium folinate
  Arms: Arm1-Methotrexate
Drug: Dactinomycin — 1.25mg/m2 (2mg max dose)intravenous every 14 days.
  Other Names: dactinomycin D
  Arms: Arm 2-Dactinomycin

SUMMARY:
The investigators conducted a randomized trial to study how well multi-day methotrexate protocol works compared to biweekly single-dose actinomycin D protocol in treating patients with low-risk gestational trophoblastic neoplasia. It is not yet known whether multi-day methotrexate protocol is as effective as biweekly single-dose actinomycin D protocol in treating patients with gestational trophoblastic neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven low-risk gestational trophoblastic neoplasia (persistent hydatidiform mole or choriocarcinoma), defined as 1 of the following:

  * Less than 10% decrease in the beta human chorionic gonadotropin (HCG) titer over 3 weekly titers
  * Greater than 20% sustained rise in beta HCG titer over two consecutive weeks
  * Histologically proven choriocarcinoma
* Stage I - III disease
* WHO risk score 0-4
* No prior chemotherapy for gestational trophoblastic neoplasia
* Signed informed consent
* Performance status - GOG 0-2
* Laboratory examination： WBC≥3.5×10(9)/L, Granulocyte count≥1.5×10(9)/L, Platelet count≥80×10(9)/L, serum bilirubin≤ 1.5 times the upper limit of normal, transaminase≤ 1.5 times the upper limit of normal, BUN, Creatinine≤ normal。 Fertile patients must use effective contraception during and for one year after study entry

Exclusion Criteria:

* Histologically confirmed placental-site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT)
* primary choriocarcinoma
* WHO risk score >4
* Previous MTX treatment for suspected ectopic pregnancy
* With severe or uncontrolled internal disease, unable to receive chemotherapy;
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Completely remission (CR) rate by single-agent | from date of treatment begin until the data serum hCG is normal for 3 consecutive weeks by single-agent chemotherapy，assessed up to 8 months
  Percentage of participants with complete response by single-agent chemotherapy. A complete response was defined as a normal hCG sustained over 3 weekly measurements.
Overall completely remission rate | from date of treatment begin until the data serum hCG is normal for 3 consecutive weeks by single-agent chemotherapy or multi-agent chemotherapy，assessed up to 12 months
  Percentage of participants with complete response by single-agent chemotherapy and those by second line multiple-drug chemotherapy after single-agent failure

SECONDARY OUTCOMES:
The duration needed to achieve complete remission after single-agent chemotherapy | from date of treatment begin until the data serum hCG is normal for 3 consecutive weeks by single-agent chemotherapy，assessed up to 8 months
  The duration needed to achieve complete remission after single-agent in two arms
The number of courses needed to achieve complete remission after single-agent chemotherapy | from date of treatment begin until the data serum hCG is normal for 3 consecutive weeks by single-agent chemotherapy，assessed up to 8 months
  The number of courses needed to achieve complete remission after single-agent chemotherapy in two arms
Incidence of Adverse Effects (Grade 3 or Higher) | through study completion, an average of 3 year
  Incidence and severity of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 in two arms
Effects on menstrual conditions and ovarian function | Prior to treatment begin，and 6 month after single-agent chemotherapy completion, an average of 2 year
  Effects on menstrual conditions and ovarian function measured by Anti-Mullerian hormone（AMH）

CONTACTS AND LOCATIONS:
Overall Officials: yang xiang, Study Director — Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiang F, Guan CL, Jiao LZ, Xu T, Wan XR, Shi SS, Wu BB, Zhang X, Zhen L, Miao JW, Tian M, Du M, Li C, Feng FZ, Yang JJ, Ren T, Zhao J, Li Y, Zhang XQ, Lu X, Xiang Y. Efficacy and safety of biweekly single-dose actinomycin D versus multiday methotrexate in low-risk gestational trophoblastic neoplasia: a prospective multicenter randomized trial. Ann Oncol. 2025 Oct;36(10):1123-1131. doi: 10.1016/j.annonc.2025.06.006. Epub 2025 Jun 19. PMID 40543844
- [Derived] Jiang F, Mao MY, Xiang Y, Lu X, Guan CL, Jiao LZ, Wan XR, Feng FZ, Ren T, Yang JJ, Zhao J. Comparing biweekly single-dose actinomycin D with multiday methotrexate therapy for low-risk gestational trophoblastic neoplasia (FIGO Score 0-4): study protocol for a prospective, multicentre, randomized trial. BMC Cancer. 2023 Aug 23;23(1):784. doi: 10.1186/s12885-023-11225-2. PMID 37612621